CLINICAL TRIAL: NCT00498043
Title: Randomized Phase II Study of Two Associations of Rituximab and Chemotherapy, With a PET -Driven Strategy, in Patients From 18 to 59 With DLBCL CD20+ Lymphoma and 2 or 3 Adverse Prognostic Factors of the Age-adjusted IPI
Brief Title: A Study of Two Associations of Rituximab and Chemotherapy, With a PET-driven Strategy, in Lymphoma
Acronym: LNH2007-3B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007.462
Record Dates: First submitted 2007-07-05; First posted 2007-07-09 (Estimated); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Lymphoma, B-Cell; Lymphoma, Large-Cell, Diffuse
Keywords: Lymphoma; PET; Chemotherapy; Rituximab
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- R-CHOP-14 (Experimental): R-CHOP14 induction regimen
  Interventions: Drug: R-CHOP14 induction regimen
- R-ACVBP14 (Experimental): R-ACVBP14 induction regimen
  Interventions: Drug: R-ACVBP14 induction regimen

INTERVENTIONS:
Drug: R-CHOP14 induction regimen — R-CHOP14 induction regimen
  Arms: R-CHOP-14
Drug: R-ACVBP14 induction regimen — R-ACVBP14 induction regimen
  Arms: R-ACVBP14

SUMMARY:
This Phase II study randomized R-ACVBP and R-CHOP as induction treatment in patients from 18 to 59 with DLBCL CD20+ lymphoma and 2 or 3 adverse prognostic factors of the age-adjusted IPI. The consolidation treatment is allocated according to the response to induction treatment assessed by PET after the 2nd and 4th induction cycles.

DETAILED DESCRIPTION:
1) Induction Arm A: 4 cycles of R-ACVBP, 2 weeks interval. After the 3rd cycle, if PET 2+ (fixing), collection of peripheral blood stem cell progenitors will be organized at the time of hematological recovery under support with G-CSF.

The consolidation treatment will depend on results of PET evaluation after cycle 2 (PET2) and cycle 4 (PET4).

* Consolidation 1A (in case of PET 2- PET 4 -):

  * High-dose Methotrexate with folinic acid rescue; 2 cycles spaced out 14 days.
  * Rituximab-Ifosfamide-Etoposide : 4 cycles spaced out 14 days
  * Cytarabine sub-cutaneous, during 4 days; 2 cycles spaced out 14 days.
* Consolidation 2 A (in case of PET 2+ PET4 -):

  * 2 cycles high-dose Methotrexate with folinic acid rescue
  * High dose with Z- BEAM conditioning regimen followed by autologous transplant.
* Salvage(in case of PET 4 +):

The patient will be treated with a salvage regimen, after a biopsy of the residual mass whenever possible.

2) Induction arm B: 4 cycles of R-CHOP, 2 weeks interval. After the 3rd cycle, if PET 2+ (fixing), collection of peripheral blood stem cell progenitors will be organized at the time of hematological recovery under support with G-CSF.

The consolidation treatment will depend on results of PET evaluation after cycle 2 (PET2) and cycle 4 (PET4).

* Consolidation 1B(in case of PET 2- PET 4 -):

  4 additional cycles of R-CHOP, 2-weeks interval
* Consolidation 2 B(in case of PET 2+ PET 4 -):

  * 2 cycles high-dose Methotrexate with folinic acid rescue
  * High dose with Z- BEAM conditioning regimen followed by autologous transplant
* Salvage(in case of PET 4 +):

The patient will be treated with a salvage regimen, after a biopsy of the residual mass whenever possible

ELIGIBILITY:
Inclusion Criteria:

* Patient with histologically proven CD20+ diffuse large B-cell lymphoma (WHO classification).
* Age from18 to 59 years, eligible for transplant.
* Patient not previously treated.
* Baseline FDG-PET Scan (PET0) performed before any treatment with at least one hypermetabolic lesion.
* Index prognostic factors (IPI) 2 or 3.
* With a minimum life expectancy of 3 months.
* Negative HIV, HBV and HCV serologies £ 4 weeks (except after vaccination).
* Having previously signed a written informed consent.

Exclusion Criteria:

* Any other histological type of lymphoma.
* Any history of treated or non-treated indolent lymphoma. However, patients not previously diagnosed and having a diffuse large B-cell lymphoma with some small cell infiltration in bone marrow or lymph node may be included.
* Central nervous system or meningeal involvement by lymphoma.
* Contra-indication to any drug contained in the chemotherapy regimens.
* Poor renal function (creatinin level >150 mmol/l), poor hepatic function (total bilirubin level >30 mmol/l, transaminases >2.5 maximum normal level) unless these abnormalities are related to the lymphoma.
* Poor bone marrow reserve as defined by neutrophils <1.5 G/l or platelets <100 G/l, unless related to bone marrow infiltration.
* Any history of cancer during the last 5 years with the exception of non-melanoma skin tumors or stage 0 (in situ)cervical carcinoma.
* Any serious active disease (according to the investigator's decision).
* Treatment with any investigational drug within 30 days before planned first cycle of chemotherapy.
* Pregnant or lactating women or women of childbearing potential not currently practicing an adequate method of contraception
* Adult patient under tutelage.
* Impossibility to performed a baseline PET scan (PET0) before randomization and treatment beginning

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 222 (Actual)
Dates: Start 2007-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Complete response rate after 4 inductive cycles with R-ACVBP14 or R-CHOP14, in DLBCL CD 20 (+) patients, presenting with 2 or 3 adverse prognostic factors of the aa-IPI Test a Pet-driven strategy Complete response rate after the 4 inductive cycles | 4 inductive cycles with R-ACVBP14 or R-CHOP14

SECONDARY OUTCOMES:
Response according to PET after 2 cycles, 4 cycles Induction toxicities Response duration Disease-, progression-, event-free and overall survival after autologous transplant Biological factors for prognosis Pharmacokinetic of rituximab | 2 cycles and 4 cycles Induction

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Coiffier, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- René Olivier Casasnovas, Dijon, France

REFERENCES:
- [Background] Casasnovas RO, Meignan M, Berriolo-Riedinger A, Bardet S, Julian A, Thieblemont C, Vera P, Bologna S, Briere J, Jais JP, Haioun C, Coiffier B, Morschhauser F; Groupe d'etude des lymphomes de l'adulte (GELA). SUVmax reduction improves early prognosis value of interim positron emission tomography scans in diffuse large B-cell lymphoma. Blood. 2011 Jul 7;118(1):37-43. doi: 10.1182/blood-2010-12-327767. Epub 2011 Apr 25. PMID 21518924
- [Derived] Girum KB, Rebaud L, Cottereau AS, Meignan M, Clerc J, Vercellino L, Casasnovas O, Morschhauser F, Thieblemont C, Buvat I. 18F-FDG PET Maximum-Intensity Projections and Artificial Intelligence: A Win-Win Combination to Easily Measure Prognostic Biomarkers in DLBCL Patients. J Nucl Med. 2022 Dec;63(12):1925-1932. doi: 10.2967/jnumed.121.263501. Epub 2022 Jun 16. PMID 35710733
- [Derived] Blanc-Durand P, Jegou S, Kanoun S, Berriolo-Riedinger A, Bodet-Milin C, Kraeber-Bodere F, Carlier T, Le Gouill S, Casasnovas RO, Meignan M, Itti E. Fully automatic segmentation of diffuse large B cell lymphoma lesions on 3D FDG-PET/CT for total metabolic tumour volume prediction using a convolutional neural network. Eur J Nucl Med Mol Imaging. 2021 May;48(5):1362-1370. doi: 10.1007/s00259-020-05080-7. Epub 2020 Oct 24. PMID 33097974
- [Derived] Tout M, Casasnovas O, Meignan M, Lamy T, Morschhauser F, Salles G, Gyan E, Haioun C, Mercier M, Feugier P, Boussetta S, Paintaud G, Ternant D, Cartron G. Rituximab exposure is influenced by baseline metabolic tumor volume and predicts outcome of DLBCL patients: a Lymphoma Study Association report. Blood. 2017 May 11;129(19):2616-2623. doi: 10.1182/blood-2016-10-744292. Epub 2017 Mar 1. PMID 28251914
- See also: Related Info — http://www.gela.org